CLINICAL TRIAL: NCT03583619
Title: A Phase II Randomized Clinical Trial of Accelerated Partial Breast Irradiation Compared With Whole Breast Irradiation With IMRT in Early Breast Cancer
Brief Title: Randomized Trial of Accelerated Partial Breast Irradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC-000498
Record Dates: First submitted 2018-06-19; First posted 2018-07-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2018-12

CONDITIONS: Breast Neoplasms; Neoplasm Recurrence, Local
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APBI (Experimental): Patients receive accelerated partial breast irradiation to tumour bed to a total dose of 40Gy, 4.0Gy per fraction, 5 fractions a week, within 2 weeks.
  Interventions: Radiation: APBI
- WBI (Active Comparator): Patients receive whole breast irradiation to a total dose of 43.5Gy, at 2.9Gy per fraction, 5 fractions a week, within 3 weeks.
  Interventions: Radiation: WBI

INTERVENTIONS:
Radiation: APBI — Patients receive radiation to the breast tumor bed to a total dose of 40Gy/10fx/2wks, using intensity-modulated radiation therapy technique.
  Arms: APBI
Radiation: WBI — Patients receive radiation to the whole breast to a total dose of 43.5Gy/15fx/3wks, using intensity-modulated radiation therapy technique.
  Arms: WBI

SUMMARY:
This study is to compare radiation toxicity of accelerated partial breast irradiation (ABPI) with whole breast irradiation (WBI) in low-risk breast cancer.

DETAILED DESCRIPTION:
This study is a single-center phase II randomized clinical trial to enroll low-risk breast cancer treat with breast-conserving surgery. All eligible patients are randomized to receive either ABPI (40Gy/10fx/2wks) or WBI(43.5Gy/15fx/3wks). Intensity modulated radiation therapy (IMRT) technique is used. Grade 2 or more acute and late toxicities are prospectively evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Life Expectation: > 5 years
* Enrollment date no more than 12 weeks after breast-conserving surgery or no more than 8 weeks after adjuvant chemotherapy
* Histologically confirmed diagnosis of invasive ductal carcinoma (grade 1-2), or mucinous carcinoma, or papillary carcinoma, or tubular carcinoma, or medullary carcinoma: primary tumor ≤ 3.0cm in maximum diameter and pN0; or histologically confirmed DCIS: primary tumor ≤ 2.5cm in maximum diameter, low-medium grade
* Unifocal tumour (confirmed by diagnostic MRI)
* No lymphovascular invasion
* ER positive (defined as medium-strongly nuclear staining in >1% of the cancer cells)
* Negative radial resection margins of >= 2 mm
* Surgical clips placed in the tumor bed
* Written informed consent.

Exclusion Criteria:

* Stage Ⅱ-Ⅲ
* Multifocal tumors
* Histologically confirmed diagnosis of invasive ductal carcinoma (grade 3), - - - invasive micropapillary carcinoma, carcinoma of lobular in situ, invasive - - - lobular carcinoma
* Paget's disease of the nipple
* Underwent oncoplastic surgery of ipsilateral breast
* Underwent neoadjuvant chemotherapy or hormonal therapy
* Previous or simultaneous contralateral breast cancer
* Undergone ipsilateral chest wall radiotherapy
* Active collagen vascular disease.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Number o participants with Grade 2 or more toxicity | 5 years
  The evaluated toxicities include the following and are evaluated by CTCAE 3.0 criteria:
  acute skin toxicity,breast swelling, breast pain,radiation pneumonitis, cardiac toxicity, pulmonary fibrosis, cosmetic result

SECONDARY OUTCOMES:
locoregional recurrence | 5 years
  ipsilateral breast and axillary nodal recurrence
overall survival | 5 years
  any death
disease-free survival | 5 years
  any recurrence or death
distant-metastasis survival | 5 years
  distant metastasis
Quality of life measured with BR-23 questionnaire | 2 years
  BR-23 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shulian Wang, M.D., Principal Investigator — National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Song YC, Sun GY, Fang H, Tang Y, Song YW, Hu C, Qi SN, Chen B, Jing H, Tang Y, Jin J, Liu YP, Lu NN, Li YX, Wang SL. Quality of Life After Partial or Whole-Breast Irradiation in Breast-Conserving Therapy for Low-Risk Breast Cancer: 1-Year Results of a Phase 2 Randomized Controlled Trial. Front Oncol. 2021 Sep 15;11:738318. doi: 10.3389/fonc.2021.738318. eCollection 2021. PMID 34604082